CLINICAL TRIAL: NCT04371861
Title: Prospective, Multi-center, Observational, Post-market Study to Assess the Safety and Procedural Success of Performing Transradial Access for Treatment of Atherosclerotic Lesions in the Lower Extremities.
Brief Title: Observational Study to Assess Transradial Access for Treatment in the Lower Extremities.
Acronym: R2P Registry
Status: Completed | Type: Observational
Sponsor: Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TIS2019-01
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Treatment of lower extremity lesion via transradial access.: Interventions performed are standard of care for treatment of a peripheral lesion.
  Interventions: Device: Peripheral Artery Treatment

INTERVENTIONS:
Device: Peripheral Artery Treatment — Peripheral lesions may be treated by any standard of care methods of treatment.

SUMMARY:
This study is designed to collect data on the complication rates and procedural success of using a transradial access approach to treat peripheral lesions in the lower extremities of a real world population.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford Category 2-5
* Subject scheduled for a transradial intervention to treat a lesion in the lower extremities.
* Willing to sign consent and agree to follow-up requirements.

Exclusion Criteria:

* Previous failed transradial access attempt
* Presence of or planned dialysis fistula.
* Planned amputation
* Previous or planned transradial access intervention +/- 30 days
* Radial artery diameter <2.5mm
* No palpable radial artery
* Established vasospastic disease
* Known allergy to contrast that cannot be managed
* Pregnant or lactating
* Mentally incompetent or a prisoner
* Currently participating in a clinical study that has not completed it's primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects planned to undergo treatment of a lower extremity lesion via transradial artery access.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Radial access site complications | Procedure
  Rates of occurrence in complications associated with transradial access.
Procedural Success | Procedure
  Successful completion of intended procedure without access complications and without conversion to femoral access.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Shishehbor, DO, Principal Investigator — University Hospitals, Cleveland, OH
Locations (8):
- United States (8):
  - UCSD, La Jolla, California
  - Northside Hospital, St. Petersburg, Florida
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Mercy Hospital, Springfield, Missouri
  - Columbia University Medical Center, New York, New York
  - Sorin Medical, Inc., New York, New York
  - University Hospitals, Cleveland, Ohio
  - Ascension Seton Hays Hospital, Kyle, Texas